CLINICAL TRIAL: NCT02368769
Title: Multidimensional Assessment of Tele-expertise for Frozen Section Diagnosis
Brief Title: Assessment of Tele-expertise for Frozen Section Diagnosis
Acronym: Télé-extempo
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Agence Regionale de Sante d'Ile de France (Other Government)
Responsible Party: Sponsor
Other Study IDs: TLM-Pathology Frozen Section
Record Dates: First submitted 2015-02-05; First posted 2015-02-23 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Frozen Sections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- During tele-expertise: Remote site interpretation of frozen section
  Interventions: Device: During Tele-expertise
- Before tele-expertise: Usual (on site) frozen section

INTERVENTIONS:
Device: During Tele-expertise
  Groups: During tele-expertise

SUMMARY:
The purpose of the study is to assess whether performing a frozen section diagnosis off site with virtual slides would be as quick and accurate as usual technique.

ELIGIBILITY:
Inclusion Criteria:

* All patients

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who need a frozen section diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 253 (Actual)
Dates: Start 2013-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Proportion of delay under 30 minutes between the sample extraction and the communication of the result to the surgeon | 30 minutes after the sample extraction

SECONDARY OUTCOMES:
Delay between extraction of the sample and the diagnosis given to the surgeon | 24h after procedure
Number of frozen section diagnosis among surgical procedures in need of frozen section diagnosis | Once a month
Overall cost of a frozen section diagnosis | 6 months after the first patient enrollment
  Sum of the durations of the professionals immobilization for performing a diagnosis x wages + costs of the telemedicine solution development and implementation.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Guettier, MD, PhD, Principal Investigator — Hôpital Bicêtre. Assistance Publique - Hôpitaux de Paris; Isabelle Durand-Zaleski, MD, PhD, Principal Investigator — DRCD URC Eco. Assistance Publique - Hôpitaux de Paris
Locations (6):
- France (6):
  - Service d'Anatomie pathologique. Hôpital Antoine Béclère, Clamart
  - Service d'anatomie pathologique. Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Service d'anatomie pathologique. Hôpital de Raincy-Montfermeil, Montfermeil
  - Service d'ORL. Hôpital du Raincy-Montfermeil, Montfermeil
  - Service d'anatomie pathologique. Hôpital Saint Antoine, Paris
  - Service de chirurgie viscérale. Hôpital des Diaconnesses, Paris

REFERENCES:
- [Background] Gould PV, Saikali S. A comparison of digitized frozen section and smear preparations for intraoperative neurotelepathology. Anal Cell Pathol (Amst). 2012;35(2):85-91. doi: 10.3233/ACP-2011-0026. PMID 22297471
- [Background] Tetu B, Fortin JP, Gagnon MP, Louahlia S. The challenges of implementing a "patient-oriented" telepathology network; the Eastern Quebec telepathology project experience. Anal Cell Pathol (Amst). 2012;35(1):11-8. doi: 10.3233/ACP-2011-0023. PMID 22233700
- [Derived] Charrier N, Zarca K, Durand-Zaleski I, Calinaud C; ARS Ile de France telemedicine group. Efficacy and cost effectiveness of telemedicine for improving access to care in the Paris region: study protocols for eight trials. BMC Health Serv Res. 2016 Feb 8;16:45. doi: 10.1186/s12913-016-1281-1. PMID 26857558